CLINICAL TRIAL: NCT04948515
Title: Association Between Gene Polymorphism of IL17 and IL 23 in Patients With COVID 19
Brief Title: Gene Polymorphism of IL17 and IL 23
Acronym: COVID 19IL17
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Saber Shafik, lecturer, Sohag University
Other Study IDs: Soh-Med-21-04-35
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples With DNA — whole blood collected on EDITA tubes for genotyping by ELISA and serum blood on plane tubes for ELISA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1 patients with severe covid 19 respiratory infections: Patients with severe covid 19 admitted to ICU, blood samples will be collected for testing different genotypes and serum level of IL 17
  Interventions: Diagnostic Test: laboratory test
- group 2 patients with non severe covid 19 respiratory infections: Patients with nonsevere covid 19 admitted to the internal ward, blood samples will be collected for testing different genotypes and serum level of IL 17
  Interventions: Diagnostic Test: laboratory test

INTERVENTIONS:
Diagnostic Test: laboratory test — genotyping of IL 17 and IL23
Diagnostic Test: laboratory test — estimation of serum level of IL 17

SUMMARY:
rates are in such considerable amount among large population base. The pathogenesis of COVID-19 implicates a potent inflammatory response, involving a complex group of mediators including interleukins. These pleiotropic cytokines are secreted at the region of inflammation and released into the circulation by a variety of different cell types, including macrophages, lymphocytes, endothelial cells, epithelial cells during sepsis and acute organ injuries. There has recently found a number of studies reporting that the cytokine storms take part in the course of COVID-19

DETAILED DESCRIPTION:
Aim Of The Study

1. To evaluate if there is an association between the IL-17, IL-23 gene polymorphism in Patients With COVID 19 by real-time PCR
2. To measure the serum level of IL17 by ELISA in COVID 19 patients by ELISA.
3. To detect if there is an association between gene polymorphism of IL17 and IL23 and severity of a condition in patients with COVID 19 Study design: a cross-sectional study.

The blood samples will be collected from patient records in COVID19 isolation hospitals in sohag governorate and isolation department in sohag university hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Covid19 positive PCR

Exclusion Criteria:

* Patients with Covid19 clinical criteria not confirmed by PCR

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: group 1 patients with covid 19 with severe infections admitted at ICU group 2 patients with covid 19 with nonsevere infections admitted at internal wards
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
genotyping of IL 17 | 3-6-2021 to 30-8-2021
  real time pcr detection of different genotypes
genotyping of IL 23 | 3-6-2021 to 30-8-2021
  real time pcr detection of different genotypes
estimation of serum level of IL 17 | 3-6-2021 to 30-8-2021
  measuring serum level of IL 17 by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: N S shafik, lecturer, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
to protect the privacy of the patient